CLINICAL TRIAL: NCT04086914
Title: Fascia Iliaca Compartment Blocks to Improve Preoperative Pain Control in Elderly Hip Fractures
Brief Title: Fascia Iliaca Compartment Blocks for Pain Control in Hip Fractures
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study withdrawn at PI's request. no patients enrolled.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00090054
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non nerve block (No Intervention): Receives no nerve block
- Nerve block (Experimental): Receives nerve block
  Interventions: Procedure: Nerve Block

INTERVENTIONS:
Procedure: Nerve Block — This group will receive a nerve block consisting of 20mL of 5mg/mL ropivicanine and 0.1mL of 10mg'mL dexamethasone.
  Arms: Nerve block

SUMMARY:
This study is comparing the use of a peripheral nerve block and standard opioid pain medications in pain control in hip fractures prior to surgery. A peripheral nerve block is a procedure that injects numbing medicine around a nerve to help decrease the pain, motion, and sensation around the painful site temporarily. The purpose of this study is to evaluate if peripheral nerve blocks are more effective for pain control than just standard opioid pain medication while decreasing the amount of side effects from opioid medication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 or older, low energy hip fracture, acute hip fracture

Exclusion Criteria:

* On anticoagulants, hardware present near injection site, preexisting nerve injury.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Mean Baseline Pain score on Visual analogue scale at initial encounter | 0-60 minutes
  pain is measured 1-10, 1 being the lowest and 10 being the highest
Mean Change from baseline pain score on the visual analogue scale | 3-8 hours after initial encounter
  pain is measured 1-10, 1 being the lowest and 10 being the highest

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043